CLINICAL TRIAL: NCT01765322
Title: Center of Assisted Reproductive Technology
Brief Title: The Effect of Laser-assisted Zona Thinning on the Implantation Rate in the Women of Advanced Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanxi Provincial Maternity and Children's Hospital (Other)
Responsible Party: Principal Investigator, Shi Wenhao, Assisted Reproductive Technology Center, Shanxi Provincial Maternity and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCHC-2013-01
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Female Urogenital Diseases
MeSH Terms: conditions — Female Urogenital Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Assisted hatching group (AH group) (Experimental): The subjects are going to participate the treatment of assisted hatching in vitro fertilization by Zona Infrared Laser Optical System (ZILOS-TK IVOS Analyzer,Hamilton Thorne Biosciences,USA).
  Interventions: Device: ZILOS-TK IVOS Analyzer
- Control group (No Intervention): The subjects are going to undergo the same procedure except for the treatment of assisted hatching.

INTERVENTIONS:
Device: ZILOS-TK IVOS Analyzer — The subjects are going to participate the treatment of assisted hatching in vitro fertilization by Zona Infrared Laser Optical System (ZILOS-TK,Hamilton Thorne Biosciences,USA)
  Arms: Assisted hatching group (AH group)

SUMMARY:
The purpose of this study is to determine whether laser-assisted zona thinning improve the implantation rate of the women of advanced age in the first IVF/ICSI cycles

DETAILED DESCRIPTION:
Registry procedures：

1. It's required to sign an informed consent form prior to the recruitment of all patients.
2. Data collection and entry need double check and supervision.

The outcome measures:

the implantation rate per embryo transfer miscarriage live birth

ELIGIBILITY:
Inclusion Criteria:

* Age: 35y ≤age≤46y
* Basal FSH value: FSH≤10IU/L
* Day-3 embryos transferred in the fresh IVF/ICSI cycles
* the number of embryos available to be transferred on Day-3: ≥one embryo

Exclusion Criteria:

* cycles with thawed/warmed embryos biopsied for PGD/PGS.
* cycles with oocyte donation transfer.
* the maximum number of previous unsuccessful IVF attempts: ≥ 3 cycles(transfer cycles)
* any cycles with the risk of OHSS, fluid in the uterine cavity, abnormal endometrium, uterine abnormalities,pelvic inflammation, and other acute maternal problems.
* One or both spouses have an abnormal karyotype (including polymorphism)

Ages: 35 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The implantation rate | 30 days
  the implantation rate per embryo in first fresh embryos transfer cycles

SECONDARY OUTCOMES:
The miscarriage | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Shi, Master, Study Director — Maternal and Children Health Care Hospital
Locations (1):
- Maternal and Children Health Care Hospital, Xi'an, Shaanxi, China